CLINICAL TRIAL: NCT00358124
Title: Insulin Glargine v Rosiglitazone as add-on Therapy in Patients Failing Sulfonylurea and Metformin Combination Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4014
Record Dates: First submitted 2006-07-28; First posted 2006-07-31 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Rosiglitazone; Metformin

INTERVENTIONS:
Drug: insulin glargine
Drug: rosiglitazone
Drug: metformin

SUMMARY:
To compare the glycemic control, as measured by HbA1C, between insulin glargine and rosiglitazone add-on therapies in patients who fail oral combination of a sulfonylurea and metformin

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of type 2 diabetes mellitus for at least one year;
* Continuous treatment with at least half maximally labeled dose of a sulfonylurea and at least 1000 mg metformin daily for at least three months ;
* Glycated hemoglobin between 7.5 and 11 % units, inclusive;
* Willingness to accept, and ability to inject insulin glargine therapy

EXCLUSION CRITERIA:

* Stroke, MI, coronary artery bypass graft, percutaneous transluminal coronary angioplasty or angina pectoris within the last 12 months;
* Congestive heart failure requiring pharmacological treatment;
* Serum creatinine > 1.5 mg/dl for males, or > 1.4 mg/dl for females;
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis;
* Planned radiological examinations requiring administration of contrasting agents;
* Clinical evidence of active liver disease, or serum ALT 2.5 times the upper limit of the normal range;
* History of hypoglycemia unawareness;
* Pregnancy or lactation;
* Failure to use adequate contraception (women of current reproductive potential only);
* Known hypersensitivity to insulin glargine, rosiglitazone or any of the components of insulin glargine rosiglitazone;
* BMI >25 kg/m2;
* Malignancy except basal cell carcinoma within the last five years;
* History of substance or alcohol abuse within last two years, or current addiction to substance or alcohol abuse;
* Any disease or condition that in the opinion of the investigator and/or sponsor may interfere with completion of the study;
* Incapability to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2001-01; Study Completion 2002-06

PRIMARY OUTCOMES:
The primary efficacy variable was the change in HbA1C from baseline to the end of therapy.
Other efficacy variables were the change from baseline in FPG, serum lipids and weight.

SECONDARY OUTCOMES:
Secondary efficacy parameters were: a mean change from baseline in FPG
Mean change from baseline in fasting insulin/C-peptide levels
Mean change from baseline in lipid levels (total cholesterol, HDL, LDL, TG, free fatty acids)
Mean change from baseline for bodyweight.
Health-related quality of life was compared between the baseline visit and the follow-up assessments

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barch, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States

REFERENCES:
- [Background] Rosenstock J, Sugimoto D, Strange P, Stewart JA, Soltes-Rak E, Dailey G. Triple therapy in type 2 diabetes: insulin glargine or rosiglitazone added to combination therapy of sulfonylurea plus metformin in insulin-naive patients. Diabetes Care. 2006 Mar;29(3):554-9. doi: 10.2337/diacare.29.03.06.dc05-0695. PMID 16505505
- [Background] Vinik AI, Zhang Q. Adding insulin glargine versus rosiglitazone: health-related quality-of-life impact in type 2 diabetes. Diabetes Care. 2007 Apr;30(4):795-800. doi: 10.2337/dc06-1712. Epub 2007 Jan 26. PMID 17259481